CLINICAL TRIAL: NCT03772990
Title: Calcium Administration in Patients Undergoing Cardiac Surgery Under Cardiopulmonary Bypass (ICARUS Trial): Prospective Randomized, Double-blind Placebo-controlled Superiority Trial
Brief Title: Calcium Administration in Cardiac Surgery
Acronym: ICARUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Collaborators: Università Vita-Salute San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21/2019
Record Dates: First submitted 2018-12-07; First posted 2018-12-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass
Keywords: inotropic support; calcium chloride; cardiopulmonary bypass; cardiac surgery
MeSH Terms: interventions — Calcium Chloride; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium chloride (Experimental): Participants randomly assigned to the experimental group will receive 15 mg/kg of calcium chloride (bolus) intravenously during separation from cardiopulmonary bypass
  Interventions: Drug: Calcium Chloride
- 0,9% Sodium Chloride (Placebo Comparator): Participants randomly assigned to the placebo group will receive equivalent amount of placebo intravenously during separation from cardiopulmonary bypass
  Interventions: Drug: 0.9% Sodium Chloride

INTERVENTIONS:
Drug: Calcium Chloride — Calcium Chloride
  Arms: Calcium chloride
Drug: 0.9% Sodium Chloride — 0.9% Sodium Chloride
  Arms: 0,9% Sodium Chloride

SUMMARY:
Termination of cardiopulmonary bypass is a critical step in any cardiac surgical procedure and requires a thorough planning. Debate about rationale of calcium administration during weaning of cardiopulmonary bypass has been conducted for several decades; however, a consensus has not been yet reached.

Perioperative hypocalcemia can develop because of haemodilution or calcium binding from heparin, albumin and citrate. Perioperative hypocalcemia is often complicated by development of arrhythmias, especially QT interval prolongation. Furthermore, low content of calcium can lead to vascular tone disorders, violation of neuromuscular transmission, altered hemostasis and heart failure, resistant to inotropic agents, especially in patients with concomitant cardiomyopathy.

On the other hand, hypercalcaemia is a dangerous complication in cardiac surgery. Among the fatal, but rather rare complications, there are acute pancreatitis and the phenomenon of the "stone heart", which is essentially a reperfusion injury of the myocardium caused by rapid calcium overload. Hypercalcaemia can also trigger rhythm disturbances, hypertension, increase systemic vascular resistance, reduce diastolic compliance and impair relaxation of the myocardium due to excessive calcium intake into the cardiomyocytes, cause coronary vasospasm and aggravate ischaemic myocardial damage, impair arterial graft blood flow during aortocoronary and mammary coronary bypass surgery.

To date, there is a lack of data indicating clinical efficacy of calcium administration before separation from CPB. Therefore, we designed this randomized controlled trial to test the hypothesis whether calcium administration at termination of CPB will reduce the need for inotropic support at the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* surgery under cardiopulmonary bypass
* valve or valve surgery + CABG
* age > 18 years
* signed informed consent

Exclusion Criteria:

* emergency surgery
* isolated aortic valve repair/replacement
* planned (before surgery) blood transfusion
* redo surgery
* known allergy to the study drug
* pregnancy
* current enrollment into another RCT (in the last 30 days)
* previous enrollment and randomization to ICARUS trial
* liver cirrhosis (Child B or C)
* transfusion during CPB
* hypo- or hyperparathyreosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 818 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2025-07-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Inotropic support | Intraoperatively
  Number of patients requiring inotropic support before transfer to intensive care unit

SECONDARY OUTCOMES:
Duration of inotropic support after surgery | 30 days after surgery
  Duration of infusion of any vasoinotropic agent at any dose
Vasoactive-inotropic score | Postoperative day 1
  Vasoactive-inotropic score will be measured on the morning of postoperative day 1. The inotropic score will be calculated using the following formula: Dobutamine dose (in mcg/kg/min) + Dopamine dose (in mcg/kg/min) + Enoximone dose (in mcg/kg/min) + [Epinephrine dose (in mcg/kg/min) x 100] + [Norepinephrine dose (in mcg/kg/min) x 100].
Plasma Ca2+ concentration before and after drug administration | Intraoperatively
Time spent in theatre after cardiopulmonary bypass | Intraoperatively
Duration of ventilation | Up to 30 day after randomization
Duration of intensive care unit stay | Up to 30 day after randomization
Myocardial infarction | Up to 30 day after randomization
  Number of patients who develop myocardial infarction
Atrial fibrillation | Up to 30 day after randomization
  Number of patients who develop postoperative atrial fibrillation
Type 1 and type 2 neurological complications | Up to 30 day after randomization
  Number of patients who develop type 1 and type 2 develop myocardial infarction
Postoperative blood loss | Postoperative day 1
  Postoperative blood (ml/kg) loss will be measured on the morning of postoperative day 1
Need for blood transfusion after surgery | Up to 30 day after randomization
  Number of patients who will need transfuion of any blood products (red cells, fresh frozen plasma, cryoprecipitate)
Intraoperative myocardial ischemia | Intraoperatively
  The presence of intraoperative myocardial ischemia will be defined during continuous intraoperative ECG monitoring after calcium chloride or placebo administration
Myocardial ischaemia on ECG after arrival to ICU | Postoperative day 1
  Number of patients who develop myocardial ischemia
Concentration of alpha-amylase after surgery | Postoperative day 1
Internal mammary artery vascular resistance (if available) | Intraoperatively
  Will be defined by intraoperative graft flow measurements

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lomivorotov, Principal Investigator — Meshalkin Research Institute of Pathology of Circulation
Locations (11):
- Sh. Mohammed Bin Khalifa Bin Salman Al-Khalifa Cardiac Center, Manama, Bahrain
- Russia (9):
  - Federal Center for Cardiovascular Surgery, Astrakhan
  - Federal Center for Cardiovascular Surgery, Chelyabinsk
  - District clinical hospital, Khanty-Mansiysk
  - B.V. Petrovsky Russian Scientific Surgery Center, Moscow
  - M. Vladimirsky Moscow Regional Research Cinical Institute (MONIKI), Moscow
  - Meshalkin Research Institute of Pathology of Circulation, Novosibirsk
  - Federal Center for Cardiovascular Surgery, Penza
  - St Petersburg University Multifunctional Clinical Centre, Saint Petersburg
  - Tomsk National Research Medical Center, Tomsk
- King Abdullah Medical City, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided